CLINICAL TRIAL: NCT06940713
Title: CONEXUS: Prospective Study of the Feasibility of Brain Connectivity Imaging by Functional Ultrasound Imaging (fUS) in Newborn Infant
Brief Title: Prospective Study of the Feasibility of Brain Connectivity Imaging by Functional Ultrasound Imaging (fUS) in Newborn Infant
Acronym: CONEXUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: C22-39; 2024-A00963-44 (Registry Identifier: ID RCB)
Record Dates: First submitted 2025-03-04; First posted 2025-04-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Neonates and Preterm Infants; Neonates or Premature Babies
Keywords: ultrasound imaging; functional ultrasound; neonatal intensive care imaging; prematurity; preterm; anoxo-ischemic encephalopathy; intrauterine growth restriction; functional connectivity; neonatology; neurodevelopment
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation | interventions — Time-Lapse Imaging; Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility of brain connectivity imaging by functional ultrasound imaging (fUS) in newborn infant (Experimental)
  Interventions: Device: Imaging Time

INTERVENTIONS:
Device: Imaging Time — fUS:
  transfontanellar functional ultrasound imaging, performed using the CONEXUS system.
  fUS-EEG:
  transfontanellar functional ultrasound imaging, performed using the CONEXUS system, performed simultaneously with an EEG examination.
  The fUS examinations consist of recording brain activity for a few minutes in one of the imaging planes (Posterior Coronal, Median Coronal, Frontal Coronal, Right Para-sagittal, Right/Left Para-sagittal, 3-plane Antero-posterior Coronal) including structures involved in brain functional connectivity networks (somatosensory, auditory, visual, salience).
  These fUS examinations are conducted to perform longitudinal follow-up of patients in the 5 different groups.
  Other Names: functional ultrasound imaging (fUS); fUS; functional ultrasound imaging combined with EEG (fUS-EEG); fUS-EEG; CONEXUS imaging

SUMMARY:
Neurodevelopmental disorders (NDD) affect how the brain develops and can lead to lifelong difficulties with movement, learning, behavior, and thinking. Every year, around one million newborns in Europe are affected by these conditions. Some babies are at higher risk of NDD due to factors such as being born extremely premature, having poor growth in the womb, experiencing a lack of oxygen at birth, or having a family history of severe NDD. However, predicting which babies will develop these disorders is currently very challenging because there are no reliable early indicators (biomarkers) to detect them.

The CONEXUS study is testing a new type of brain imaging technology called functional ultrasound imaging (fUS) to see if it can help assess brain function in newborns at high risk of NDD. This technique measures brain activity by detecting small changes in blood flow, similar to an ultrasound scan but using advanced imaging technology. Researchers believe this method, known as fC-fUS imaging, could help identify early signs of neurodevelopmental disorders.

Preliminary studies have shown that fUS imaging can detect brain activity changes in newborns, such as differences between sleep states or during epileptic seizures. The CONEXUS study will expand on this by improving the imaging technology and testing it in a larger group of newborns, including those born prematurely, those with restricted growth, those who needed cooling treatment after birth due to lack of oxygen, and those at risk for autism spectrum disorder (ASD).

The study is being conducted in multiple hospitals in France over five years, involving newborn intensive care, pediatrics, and child psychiatry teams. It is a feasibility study, meaning researchers aim to test whether this imaging technique is practical and effective for use in newborns. Babies will have short, painless fUS scans that focus on brain regions involved in movement, hearing, vision, and attention.

Ultimately, the goal of CONEXUS is to demonstrate that fC-fUS imaging can help doctors understand early brain development and identify signs of neurodevelopmental disorders before symptoms appear. If successful, this technique could improve early diagnosis, allowing doctors to start treatment sooner and improve long-term outcomes for affected children. This research has the potential to transform neonatal care by providing a new tool for detecting and monitoring brain function in newborns.

DETAILED DESCRIPTION:
Introduction

Neurodevelopmental disorders (NDD) result from an alteration in brain development and represent a major public health problem, affecting 1 million newborns in Europe each year. Neurodevelopmental disorders are the source of permanent disabilities that manifest as motor, cognitive, learning, or behavioral dysfunction. Prenatal or neonatal factors considered high risk for NDD include: extreme prematurity, newborns with intrauterine growth retardation, brain growth abnormalities, anoxic-ischemic encephalopathy (AIE) with an indication for therapeutic hypothermia, and a family history of severe NDD in the first degree. Establishing a reliable prognosis for neurodevelopmental disorders is extremely difficult because there are currently no early biomarkers to detect and assess potential long-term deficiencies.

The CONEXUS protocol aims to evaluate whether a unique neuroimager, using ultrafast ultrasound imaging, is capable of assessing, at the patient's bedside, the brain's functional connectivity (fC) in newborns at high risk of NDD. This neuroimager uses functional ultrasound imaging (fUS), a technique developed within the Physics for Medicine laboratory (Paris), and thus constitutes the central medical device of this protocol.

Device

The CONEXUS system is composed of several elements necessary for functional brain imaging of newborns: the Conexus station (similar to an ultrasound machine) on which the Conexus software is installed (allowing the acquisition and processing of ultrasound data necessary for imaging), the ultrasound probe (a physical element allowing the emission and reception of ultrasounds, similar to an ultrasound probe), and the headset (a small system adapted to the anatomy of the patient's head and allowing the probe to be held in place over the fontanelle).

This system allows mapping of brain activity via subtle changes in cerebral blood volume. It is quite similar to an ultrasound machine but uses different image reconstruction and signal processing techniques, which give it its properties. Our research hypothesis: the evaluation of fC by fUS imaging (fC-fUS imaging) is feasible in newborns and could eventually reveal early biomarkers of perinatal brain diseases.

This hypothesis is supported by our preliminary work on neonatal fUS imaging: we have shown the possibility of performing fUS imaging in some newborns and thus measuring a change in brain activity during sleep state changes or during epileptic seizures, as well as at different stages of neurodevelopment (premature vs. term). The CONEXUS study aims to go further thanks to improved technical capabilities and ergonomics (notably the ultrasound probe) allowing multiplane imaging approaching 3D imaging and imaging a large clinical cohort including different stages of development and various pathological risks (term newborns, premature newborns, newborns with intrauterine growth retardation (IUGR), AIE newborns placed in therapeutic hypothermia, and newborns at risk of autism spectrum disorder (ASD)).

Study

Conexus is a descriptive research study of neonatal brain connectivity using fUS imaging. It is a national clinical investigation involving the Neonatal Intensive Care and Pediatrics/Maternity and Child Psychiatry Services of the Robert Debré Hospital, and concerning a medical device (MD), classified as IIa non-CE marked, without the objective of establishing CE marking (IC 4.4). It therefore uses a new medical device for research purposes, the "Conexus" system, which is a joint production of the Physics for Medicine Paris laboratory and the Iconeus company carried out under a scientific collaboration contract. It is a prospective feasibility pilot study, multicentric, open, controlled, and non-randomized. The research will last 5 years, including 3 years of inclusion.

The fUS examinations consist of recording brain activity for a few minutes in one of the imaging planes (Posterior Coronal, Median Coronal, Frontal Coronal, Right Para-sagittal, Right/Left Para-sagittal, 3-plane Antero-posterior Coronal) including structures involved in brain functional connectivity networks (somatosensory, auditory, visual, salience). These fUS examinations are conducted to perform longitudinal follow-up of patients in the different groups.

CONEXUS aims to prove the potential of fC-fUS to characterize and monitor brain functions, understand the developing brain, and search for biomarkers of neurological deficiencies. The definition of early biomarkers of neurodevelopmental disorders would allow early management to guide therapeutic decisions and improve treatment effects. fUS imaging and fC-fUS evaluation have the potential to transform the clinical management of newborns and address a pressing clinical need in neonatology.

Objectives

Main objective: To evaluate the feasibility of acquiring data via fUS imaging of brain functional connectivity in 4 groups (G1 to G4) of newborns at high risk of NDD and a control group of term newborns (G5): group G1 of premature newborns born before 32 weeks of amenorrhea (WA) (N = 26), group G2 of newborns with anoxic-ischemic neonatal encephalopathy >36 WA (AIE) (N = 10), group G3 of newborns with IUGR <10th percentile (N = 10), group G4 of newborns from siblings with autism spectrum disorder (ASD) (N = 10), compared to a control group (G5) of term newborns without neurological pathology (N = 20).

Secondary objectives:

* To study the evolution of fUS connectivity in premature infants (G1), from birth to corrected term in relation to brain functional connectivity in term newborns (G5), newborns with anoxic-ischemic encephalopathy (AIE) (treated with therapeutic hypothermia) (G2), newborns with IUGR (G3), and newborns from siblings with at least one child with autism spectrum disorder (ASD) (G4).
* To identify a posteriori within the groups of premature infants (group G1), newborns with AIE (group G2), newborns with IUGR (group G3), and newborns from siblings with ASD (group G4), any early markers of an abnormal neurodevelopmental trajectory (identified based on neuropsychological evaluation at 2 years).
* To create 3D vascular atlases specific to fUS imaging to document the evolution of cerebrovascular structures (vessels >100µm) in premature infants (group G1), newborns with AIE (G2), newborns with IUGR (G3), and term newborns (group G5), as these data are currently non-existent.
* To create for the first time simultaneous clinical fUS-EEG recordings to study their possible correlations for the 5 groups. By studying possible correlations, we mean, for example, the study of the possible difference in the nature of fUS signals during clearly identified EEG activity periods (e.g., sleep phases).

ELIGIBILITY:
Inclusion Criteria:

1. For group G1 (Premature babies):

Gestational children:

1a. Between 23 WA+5 days and 27 WA +6 days (extremely preterm) (G1) or

1b. Between 28 WA+0 days and 31 WA+6 days (very preterm) (G1)

2. For the G2 group (AIE):

* Children of gestational age> 36 WA + 0 days
* with neonatal anoxo-ischemic encephalopathy
* treated with controlled therapeutic hypothermia (group G2)

  3. For the G3 Group (IUGR): Gestational age between 32 WA+0 days and 40 WA+6 days and with IUGR intrauterine growth restriction: birth weight < 10 p and/or head circumference < 10 percentile (G3 group);

  4. For the G4 group :
* Siblings with at least one child with signs of autism spectrum disorder
* less than 6 months of age at baseline (G4 group)

  5. For the G5 group (control):
* Children of gestational age between 39 WA and 40 WA + 6 days
* without pathology during pregnancy (no vasculoplacental pathology, no threat of premature delivery, no maternal corticosteroid therapy, no consumption of toxic substances)
* at birth: Apgar greater than 6 at M10; pH>7.20; lactate< 6 mmol/l; eutrophic; Birth weight >10p; Cranial Perimeter >10p

  6. Consent of the holders of parental authority 7. Child affiliated to or in receipt of a social security scheme

Exclusion Criteria:

* Person subject to a judicial safeguard measure (guardianship, curatorship or safeguard of justice)
* Known malformative pathology;
* Known chromosomal abnormality;
* Known allergy to silicone

Max Age: 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of acquiring quantitative brain functional connectivity assessment using fUS data in 4 groups (G1 to G4) of newborns at high risk of neurodevelopmental disorder and a control group of term newborns. | up to 16 weeks
  Each fUS acquisition, for each patient, each acquisition time point, each imaging plane, consists of a succession of fUS images recorded over a duration ranging from 5 to 10 minutes. The acquisition will be considered successful if at least 50% of the fUS images do not show motion artifacts (criterion used in our preliminary studies) (validity criterion) and if vascular structures are visible at a depth >50% of the maximum depth (sensitivity criterion). If these two criteria are met, we can then average the fUS signal over the functional areas and calculate a correlation matrix.

SECONDARY OUTCOMES:
Feasibility of longitudinal quantification of fUS connectivity of preterm (from birth to equivalent term age) and term newborns in different connectivity networks | up to 16 weeks
  Static connectivity matrices are calculated for specific imaging planes via signals averaged over predefined functional areas (including: thalamus, precentral gyrus, postcentral gyrus, temporal lobe, Heschl's gyrus, insula, anterior and posterior cingulate cortex, frontal lobe, striatum, amygdala, visual cortex V1 V2) within an fUS acquisition. These matrices are compared after Fisher transformation via an ANOVA (Analysis of variance) and post hoc student test with correction (significance levels 95%)
Potential correlation between fUS connectivity assessment and neuropsychological assessment at 2 years within the groups of newborns at high risk of neurodevelopmental disorder | 2 years
  Quantitative connectivity assessment of the preterm newborn group will be compared to the Brunet-Lézine neurodevelopmental score at 2 years, to identify a potential correlation.
Feasibility of acquisition of 3D vascular atlases specific to fUS imaging in order to document the evolution of cerebrovascular structures in newborns at high risk of neurodevelopmental disorder and term newborns | up to 16 weeks
  No statistical analysis and no quantitative metrics, the measurement is of documentary value.
Quantify potential correlates between fUS and EEG data thanks to the simultaneous fUS-EEG clinical recordings in newborns at high risk of neurodevelopmental disorder and term newborns. | up to 16 weeks
  Comparison of connectivity between different sleep phases. The occurrences of different connectivity states will be evaluated for each group in the two sleep phases and tested via an ANOVA and post hoc Tukey's test, as for secondary outcome measure 2.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie BIRAN, MD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France